CLINICAL TRIAL: NCT04224805
Title: Evaluation of the Use of Bone-borne CAD/CAM Surgical Guides in Orthognathic Surgery Cases Requiring Le Fort I Osteotomy
Brief Title: The Use of Bone-borne Guides in Orthognathic Surgery Cases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Haitham Mohammed Abou Eleneen, Assistant lecturer of Oral and Maxillofacial Surgery, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AlexandriaU- FacDentistry
Record Dates: First submitted 2020-01-07; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Dentofacial Deformities
Keywords: Le Fort; Orthognathic surgery; Virtual surgical planning
MeSH Terms: conditions — Dentofacial Deformities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Interocclusal conventional splint is used to reposition the maxilla.
  Interventions: Device: 3D interocclusal conventional splint
- Study (Experimental): Bone-borne splint is used to reposition the maxilla.
  Interventions: Device: Bone-borne CAD/CAM splint

INTERVENTIONS:
Device: Bone-borne CAD/CAM splint — 3D printed splint that repositions the maxilla with the zygomatic buttress as a reference.
  Arms: Study
Device: 3D interocclusal conventional splint — Interocclusal splint that relies on the centric relation of the condyle as well as occlusion.
  Arms: Control

SUMMARY:
The present study was conducted to evaluate a new design of the intermediate stent that is used in orthognathic surgery cases requiring Le Fort I osteotomy. The new design relied on referencing the maxillary segment to the zygomatic buttress. The study was carried out as a randomized controlled clinical trial in which 16 patients were enrolled according to the inclusion and exclusion criteria. In control group (n=8) conventional interocclusal splint was used and in study group (n=8) the proposed intermediate stent was used.

DETAILED DESCRIPTION:
Background: Dentofacial deformities have many negative consequences in the form and function of head and neck region. This includes breathing, swallowing, speech and temporomandibular disorders. It is estimated that in about 19% of orthodontic patients, orthognathic surgery is required along with the orthodontic procedure. The introduction of CAD/CAM technology in orthognathic surgery planning has facilitated the procedure and allowed for more predicted results. Aim of this study: The aim of the present study is to propose a new design of the intermediate stent that relates the mobilized maxilla to a fixed anatomical landmark in the skull which would allow for more accurate positioning of the maxilla during orthognathic surgery. Materials and methods: This study was conducted on sixteen patients who have been undergone Le Fort I osteotomy procedure. Eight of them (group A) were treated via a conventional stent while the other eight patients (group B) via a CAD/CAM bone-borne stent. Postoperative patient evaluation was performed by comparing the predicted maxillary position to the resultant position postoperatively. This was done via 3D reconstruction CT scans.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dentofacial deformity requiring Le Fort I osteotomy

Exclusion Criteria:

* Patients with severe asymmetry

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Error of superimposition | 2 weeks
  Superimposition error between planned and actual maxillary position

SECONDARY OUTCOMES:
Visual Analogue Scale | 3 months
  Pain assessed by score from 0 to 10 with 0 no pain and 10 severe unbearable pain.
Procedure duration | 1 day
  Time of the surgery using the splint

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt